CLINICAL TRIAL: NCT06107270
Title: Effect of Deep Neck Flexors Biofeedback Training and Post Isometric Relaxation in Chronic Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohammed Hamed Sherif, Effect of Deep Neck Flexors Biofeedback Training and Post Isometric Relaxation in Chronic Mechanical Neck Pain, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNFT+PIR technique
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Deep Neck Flexors Training; Post Isometric Relaxation

STUDY DESIGN:
Intervention Model Description: Group A (n=15) will be treated by Post Isometric Relaxation, infrared radiation and continuous ultrasound for 12 sessions (3 sessions per week for four weeks).
  Group B (n=15) will be treated by DNF training, infrared radiation and continuous ultrasound for 12 sessions (3 sessions per week for four weeks) Group C (n=15) will be treated by Post Isometric Relaxation combined DNF training, infrared radiation and continuous ultrasound for 12 sessions (3 sessions per week for four weeks)
Who Masked: Participant, Outcomes Assessor
Masking Description: All the patients will be blinded to group allocation by ensuring that they were unaware of the exercise performed by the other group. To maintain the blinding, the intervention sessions will be delivered separately to members of each treatment group, The allocation will be conducted by another researcher before the baseline.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): (n=15) will be treated by Post Isometric Relaxation, infrared radiation and continuous ultrasound for 12 sessions (3 sessions per week for four weeks).
  Interventions: Device: therapeutic ultra sound; Device: infra red radiation; Other: post isometric relaxation
- Group B (Experimental): (n=15) will be treated by DNF training, infrared radiation and continuous ultrasound for 12 sessions (3 sessions per week for four weeks)
  Interventions: Device: pressure biofeedback; Device: therapeutic ultra sound; Device: infra red radiation
- Group C (Experimental): (n=15) will be treated by Post Isometric Relaxation combined DNF training, infrared radiation and continuous ultrasound for 12 sessions (3 sessions per week for four weeks)
  Interventions: Device: pressure biofeedback; Device: therapeutic ultra sound; Device: infra red radiation; Other: post isometric relaxation

INTERVENTIONS:
Device: pressure biofeedback — uninﬂated pressure sensor will be kept below the neck suboccipital
  Arms: Group B; Group C
Device: therapeutic ultra sound — continuous US waves of 1 MHz frequency and 1-1.5 W/cm2 power
Device: infra red radiation — (R 125, 250watt, Philips)
Other: post isometric relaxation — sustained contraction followed by relaxation
  Arms: Group A; Group C

SUMMARY:
This study will be conducted to explore the superiority of effectiveness between Muscle energy technique combined with Deep Neck Flexors training, MET alone, or DNF training alone in terms of pain intensity, neck function, forward head posture, cervical range of motion and Deep Neck Flexors Muscles endurance in patients with chronic mechanical neck pain(CMNP).

DETAILED DESCRIPTION:
Patients will be grouped into three groups; each group composed of 15 patients suffering from CMNP. The personal history of each patient who participated in the study will be collected, the patient will receive an oral explanation of the procedures and signed a consent form . The weight and height of each patient will be obtained using the standard weight scale. The pain intensity level will be assessed via a visual analogue scale (VAS). The disability level will be assessed via neck disability index (NDI). The forward head posture will be assessed via photographic method of Craniovertebral angle (CVA) and the angle will be calculated by using kinovea software. The range of motion will be assessed via universal goniometer (UG). The endurance of the neck muscles will be assessed via pressure biofeedback unit (PBU). Assessment will be done before treatment and after 12 treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 20-40 years of female and male patient.
2. Patient with neck pain duration more than 3 months and less than one year.
3. Subjects who could not maintain blood pressure at increments of 24 mmHg from the initial 20 mm Hg
4. Patients who have moderate neck pain and disability scoring 15 to 24 from 50 on neck disability index. .
5. Pain intensity more than 3 and less than 7 on visual analogue scale (VAS)
6. CVA less than 49°

Exclusion Criteria:

1. People with severe neck pain. (Disability scoring more than 25 on Neck Disability Index)
2. If they are participated in a neck rehabilitation program over the last 6 months
3. Major circulatory or respiratory disorder
4. Pregnant women or 3 months postnatal
5. Patient with structural instability and degenerative conditions of cervical spine.
6. Body Mass Index more than 30.
7. Post traumatic or infective conditions.
8. Any surgeries around cervical spine
9. Vertigo patient
10. Un-cooperative patient (Gupta et al., 2022).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
pain severity | 4 weeks
  Visual Analogue Scale It is a 10 cm or 100 mm psychometric response scale to measure pain intensity based on numerical values, anchored by a score of 0 no pain and score 10 worst pain The patient will be asked to place a horizontal mark on the continuous 10 cm line in which they could feel. A ruler will be then used to measure the distance from zero and the recorded number will be rounded to the nearest number Visual Analogue Scale .It is a 10 cm or 100 mm anchored by a score of 0 no pain and score 10 worst pain
functional disability | 4 weeks
  Neck Disability Index . 0% means no activity limitation, and 50 points or 100% means complete activity limitation
Deep Neck Flexors muscle endurance | 4 weeks
  Pressure biofeedback unit . used for muscular assessment of longus colli and longus capitus.

SECONDARY OUTCOMES:
craniovertebral angle (CVA) | 4 weeks
  Kinovea (version 0.9.5) will be used to calculate the CVA
cervical range of motion | 4 weeks
  Universal goniometer.to measure the active cervical range of motion in all directions.

IPD SHARING:
Plan to Share IPD: No